CLINICAL TRIAL: NCT06846372
Title: Effect of 3D Integration of Facial Scanning, Intraoral Scanning and CBCT on Patient Satisfaction and Occlusion of Temporary and Permanent Full Arch Implant Supported Prosthesis
Brief Title: 3D Integration of Facial , Intraoral Scanning and CBCT on Patient Satisfaction and Occlusion of Temporary, Permanent Implant Supported Prosthesis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A04012023RP
Record Dates: First submitted 2024-11-22; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-02

CONDITIONS: Occlusal Analysis; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Temporary full arch implant supported prosthesis. (Active Comparator): full arch temporary implant supported prosthesis will be fabricated for the first group using PMMA material
  Interventions: Device: occluscence; Other: patient satisfaction
- permanent full arch implant supported prosthesis. (Active Comparator): Permanent full arch implant supported prosthesis will be fabricated for the second group from zirconia
  Interventions: Device: occluscence; Other: patient satisfaction

INTERVENTIONS:
Device: occluscence — The OccluSense handheld is a battery powered device which uses your local wireless network to transmit the recorded data to the OccluSense-iPad-App.
  The inductive charger provides wireless power transfer. Fully charged batteries allow up to 4 hours usage of the device.
Other: patient satisfaction — • patient satisfaction will be evaluated by using (VAS score) on a line from 0 to 100mm (0 mm is very bad /100 mm is excellent).
  Are you satisfied with the esthetic outcome of the treatment? Does the treatment answer to your expectations? Would you choose the same treatment again? Is your ability to chew improved after placement of the implant prothesis? Did you find the complete treatment time too prolonged?

SUMMARY:
This study will aim to evaluate the effect of complete digital workflow for construction of temporary and permanent full arch implant supported screw retained restoration by the 3D integration of facial scanning, intraoral scanning and CBCT regarding patient satisfaction (VAS score) and occlusion.

DETAILED DESCRIPTION:
Aim: evaluating the effect of complete digital workflow for construction of temporary and permanent full arch implant supported screw retained restoration by the 3D integration of facial scanning, intraoral scanning and CBCT regarding patient satisfaction (VAS score) and occlusion.

Methods:1. Four radio opaque markers on patient's face will be placed. The first facial scan will be done (FS1) using a facial scanner (Bellus3D mobile application) while the patient is smiling.

2.A proper size of triple tray will be selected and adjusted if needed, and the impression material will be kept to the minimum required to avoid any overextension that can cause forced soft tissue displacement. The handle will be removed and 3 markers will be placed on the front of the triple tray.

3- The tray will be filled with heavy body vinylpolysiloxane (VPS) material and inserted in patient's mouth. The patient will be instructed to close in habitual occlusion and the second facial scan (FS2) will be taken with the head in the same position.

4. Both facial scans will be imported to a dental software design program as STL1 and STL2 files, respectively. A CBCT will be taken while the markers are still in place. Through the face scans and CBCT scan, make sure the patient is in a natural head position where reference lines (Frankfurt plane and occlusal plane) are confirmed to be parallel to the floor. The patient will be instructed to stay still.

5. The maxillary and mandibular intraoral scans will be taken with jaw relation record (STL3) using an intraoral scanner and scan the triple tray on both sides and external borders with markers in place using the Bio copy tool in Prime scan (STL4).

6. All scans will be exported to the design software. and use the design module of CAD software to superimpose the facial scans (STL1 and STL2) by using markers as reference points 7.The intraoral scans will be integrated to facial scans by using the inter arch impression STL4 (Scan of triple tray or Bio copy) as a merging tool. Complete the facially generated diagnostic wax up (STL5).

8. The completed maxillary diagnostic wax up (STL5) will be exported, pre op intraoral scans (STL3) and will be imported to implant planning software using STL markers to merge STL files correctly. the STL files with CBCT will be merged, and the interim restoration will be designed in the software program and it will be 3D printed.

9.the interim restoration will be inserted and the patient satisfaction and occlusion will be evaluated.

10. The patient will receive postoperative instructions until the definitive prostheses will be fabricated.

11.After insertion of the permanent restoration the patient satisfaction and occlusion will be evaluated.

Evaluation:• Occlusal analysis will be evaluated by occluo-scence (measuring the balance of occlusal contact forces, the sequence, strength, and density of the occlusal contacts The patient's recorded occlusal information will be transmitted and displayed on the app.

• patient satisfaction will be evaluated by using (VAS score) on a line from 0 to 100mm (0 mm is very bad /100 mm is excellent).

Are you satisfied with the esthetic outcome of the treatment? Does the treatment answer to your expectations? Would you choose the same treatment again? Is your ability to chew improved after placement of the implant prothesis? Did you find the complete treatment time too prolonged?

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals with the completely edentulous maxilla and mandible rehabilitated by six implants.

Exclusion Criteria:

* individuals with uncontrolled systemic diseases that affect the success of implant survival rate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
occlusion of temporary and permanent full arch implant supported prosthesis constructed by digital workflow | "through study completion, an average of 1 year"

SECONDARY OUTCOMES:
patient satisfaction of temporary and permanent full arch implant supported prosthesis constructed by digital workflow using (vas score) | "through study completion, an average of 1 year"
  • patient satisfaction will be evaluated by using (VAS score) on a line from 0 to 100mm (0 mm is very bad /100 mm is excellent).
  Are you satisfied with the esthetic outcome of the treatment? Does the treatment answer to your expectations? Would you choose the same treatment again? Is your ability to chew improved after placement of the implant prothesis? Did you find the complete treatment time too prolonged?

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Abdo El Syad, Professor, Principal Investigator — faculty of dentistry Mansoura university
Locations (1):
- Faculty of dentistry Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhlman DC, Almuzian M, Coppini C, Alzoubi EE. Accuracy (trueness and precision) of four tablet-based applications for three-dimensional facial scanning: An in-vitro study. J Dent. 2023 Aug;135:104533. doi: 10.1016/j.jdent.2023.104533. Epub 2023 May 4. PMID 37149254